CLINICAL TRIAL: NCT00264433
Title: An Open-Label Phase 2a Study in Subjects With N-Cadherin Positive, Advanced or Recurrent Solid Tumors to Investigate the Safety and Efficacy of ADH-1 Administered Intravenously as a Single Agent (Adherex Protocol Number AHX-01-201)
Brief Title: A Study of the Safety and Effects of ADH-1 Given Intravenously as a Single Agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adherex Technologies, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adherex Protocol # AHX-01-201
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2007-08-06 (Estimated); Status verified 2007-08

CONDITIONS: Neoplasms
Keywords: Cancer; Tumors; Neoplasms; Anticarcinogenic Agents; Antineoplastic Agents; Cadherins; Non-Small-Cell Lung Carcinoma; Esophageal Cancer; Gastric Cancer; Renal Cell Carcinoma; Hepatocellular Carcinoma; Adrenocortical Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Adrenocortical Carcinoma | interventions — N-Ac-CHAVC-NH2

INTERVENTIONS:
Drug: ADH -1 (Exherin™)

SUMMARY:
N-cadherin, a protein involved in blood vessel cell binding, is increased as cancer progresses, and is on the surface of many tumor cells. ADH-1 blocks N-cadherin. This study will test the safety and effects of ADH-1 in subjects with specific incurable, solid tumors with a protein biomarker called N-cadherin. This study will examine the clinical activity of ADH-1.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male and female patients > or = 18 years of age with a solid tumor(s) refractory to standard curative therapy or for which no curative therapy exists
* Histologically proven advanced and/or metastatic solid tumor of one of the following histologies:

  * non-small cell lung cancer (squamous or non-squamous histology),
  * gastroesophageal carcinoma (squamous or adenocarcinoma histology),
  * renal cell carcinoma,
  * hepatocellular carcinoma,
  * adrenocortical carcinoma
* Measurable disease
* Immunohistochemical evidence of N-cadherin expression (at least 1+ positive) in archived or fresh tumor tissue
* Adequate performance status and organ function, as evidenced by hematological and biochemical blood testing and electrocardiogram (ECG)

Exclusion Criteria:

* Receipt of ADH-1 prior to this clinical study
* Chemotherapy, radiotherapy, or any other investigational drug within 30 days before study entry
* History of spinal cord compression, or history of primary brain tumor(s) or brain metastases (known or suspected) unless any lesions have completely resolved following appropriate treatment and there has been no recurrence for at least 6 months
* History of tumors that have shown clinically significant evidence of active bleeding (e.g., gross hemoptysis, hematemesis, hematuria, melena, or bleeding superficial tumor) within 12 weeks before study entry
* Stroke, major surgery, or other major tissue injury within 30 days before study entry
* History of:

  * uncontrolled congestive heart failure,
  * coronary artery disease, or life threatening arrhythmias;
  * myocardial infarction less than 12 months prior to study entry;
  * significant ECG abnormalities; or
  * known hypercoagulable states

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Florida Cancer Specialist, Fort Myers, Florida
  - Lineberger Comprensive Cancer Center, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Centre, Durham, North Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Centre for Clinical Research, Halifax, Nova Scotia
  - The Ottawa Hospital Regional Cancer Center (TOHRCC), Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Jewish General Hospital, Montreal, Quebec

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com